CLINICAL TRIAL: NCT06357871
Title: Role of Renal Biopsy in the Suspicion of Nephrotoxicity of Immunotherapy (Checkpoint Inhibitors) in Solid Cancer
Acronym: NEPHROTOX
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: University Hospital, Strasbourg, France (Other); CHU de Reims (Other); Centre Hospitalier Régional Metz-Thionville (Other); European Georges Pompidou Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2023PI178
Record Dates: First submitted 2024-04-05; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2023-11

CONDITIONS: Chemotherapeutic Toxicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Test cohort: To establish the score
  Interventions: Other: No intervention
- Validation cohort: To validate the score
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Checkpoint inhibitors represent a new class of widely used immunotherapy, however with immune-mediated adverse effects, with renal damage estimated at 1.4% and 4.9% depending on the series.

Acute tubulointerstitial nephritis (ATNI) represents the most common type of damage, although there are other types of damage, associated or not with NTIA.

We aim to establish a probability score for the presence of histological NTIA lesions in a patient treated with CPI who presents with acute renal failure in order to guide the nephrologist and oncologist in their management in the event of AKI at the CPI, and determine the usefulness of a PBR to guide the suspension/resumption of immunotherapy +/- associated corticosteroid therapy; avoiding a PBR exposing to a high iatrogenic risk and sometimes impossible.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old Diagnosis of solid cancer treated by immunotherapy such as checkpoint inhibitor, associated or not with chemotherapy Renal failure having benefited from a renal biopsy

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include all patients hospitalized for kidney biopsy in the context of acute renal failure with CPI treatment.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Estimation using a multivariate model of the factors associated with the histological presence of NTIA vs NTA lesions in a patient treated with CPI | between January 2020 and December 2024

CONTACTS AND LOCATIONS:
Overall Officials: Adrien Flahault, MD, PhD, Principal Investigator — CHRU de Nancy
Locations (1):
- CHRU de Nancy, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No